CLINICAL TRIAL: NCT00941538
Title: A Cluster Randomized Controlled Screening Trial for Nasopharyngeal Carcinoma in Southern China (CRCSTNPC Study)
Brief Title: Cluster Randomized Controlled Screening Trial for NPC
Acronym: CRCSTNPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Research Institute of Zhongshan City (Other Government); Sihui Cancer Institute (Other)
Responsible Party: Principal Investigator, Hong Ming-huang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CRCSTNPC
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Nasopharyngeal Cancer; Screening; Morality
Keywords: nasopharyngeal cancer; screening; early detection; mortality; randomized control trial; Epstain-Barr Virus
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Residents aged 30-69 years in eight screening towns in the intervention group are invited to screening marker tests - IgA antibodies to EBV VCA/IgA and EBV nuclear antigen-1 (EBNA1/IgA) by ELISA.
  The trial will use two minimally acceptable false-positive rates (i.e., 10% and 3%) as the cutoffs to define "medium-risk" (seropositive, 0.65 ≤ score < 0.98) and "high-risk" participants (seropositive, score ≥ 0.98). After a blood test, participants whose EBV-based risk exceeds the predefined "high-risk" threshold (score ≥ 0.98) will be referred to endoscopy for clinical evaluation. Participants who are defined as "medium-risk" or "high-risk" (score ≥ 0.65) will be followed annually through blood testing and linkage to registers. The remaining participants (seronegative, score < 0.65) will be asked to return for a follow-up visit after five years.
  Interventions: Diagnostic Test: Experimental: Screening with EBV VCA/EBNA1-IgA testing
- Control (No Intervention): The individuals aged 30-69 in the other eight towns will be included as controls, which is a comparable population that will not be screened for NPC.

INTERVENTIONS:
Diagnostic Test: Experimental: Screening with EBV VCA/EBNA1-IgA testing — Participants in the screening towns will be offered screening tests. Those with high-risk scores will be referred to a diagnostic workup examination using fiberoptic endoscopy examination and nasopharyngeal biopsies if suspicious lesions is observed.
  Other Names: Diagnostic work-up using fiberoptic endoscopy examination and/or nasopharyngeal biopsies
  Arms: intervention

SUMMARY:
This study is aimed to estimate the effectiveness of an Epstein-Barr virus (EBV) serology-based screening program to reduce nasopharyngeal carcinoma (NPC) mortality in a cluster randomized controlled trial in an NPC high-risk population. Sixteen towns in Sihui and Zhongshan Cities, China will be selected, with eight allocated to the screening group and eight to the control group. Cantonese residents aged 30-69 years with no history of NPC will be included. Residents in the screening towns will be invited to undergo serum EBV VCA/EBNA1 IgA antibody tests.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) has a high prevalence in southern China. Sihui and Zhongshan cities are located along the Pearl River in Guangdong Province, China, and are well known for a high incidence of NPC worldwide. During the last 20 years, Screening for NPC has been demonstrated to increase the early detection rate of NPC in endemic regions. It is well shown that the effect of Epstein-Barr virus (EBV) serological antibodies is elevated several years before NPC diagnosis; therefore, EBV antibodies have been considered screening markers for NPC. However, none of the studies have reported the impact of screening on NPC-specific mortality.

This study aims to launch a cluster-randomized screening trial with combined VCA/IgA and EBNA1/IgA measurement by ELISA as the primary screening method in these 2 cities to examine the impact of EBV serological screening on NPC-specific mortality. Residents aged 30-69 years in eight screening towns in the intervention group will be invited to EBV antibody tests-IgA antibodies to EBV VCA/IgA and EBV nuclear antigen-1 (EBNA1/IgA) by ELISA. The primary objective of this trial is to assess an estimate of the EBV serological antibody-based screening for NPC on NPC-specific in the populations with a high incidence of NPC

ELIGIBILITY:
Clusters

1. Inclusion criteria 1) the town located in Sihui or Zhongshan city; 2) the town established a tertiary cancer prevention network; 3) the medical staff in the town hospitals agreed to take part in.
2. Exclusion criteria 1) having conducted NPC screening program.

Individuals

1. Inclusion criteria 1) being aged 30-69 years; 2) being Cantonese; 3) having signed the informed consent; 4) having an Eastern Cooperative Oncology Group score of 0-2; and 5) having a good physical or psychological condition and consciousness.
2. Exclusion criteria 1) having prevalent NPC.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87600 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate of NPC at 12 years by intervention group | December, 2019
  NPC mortality rate will be compared between screening group and control group at 12-year follow-up.

SECONDARY OUTCOMES:
All-cause mortality at 12 years by intervention group | December, 2019
  All-cause mortality rate will be compared between screening group and control group at 12-year follow-up.
NPC incidence at 12 years by intervention group | December, 2019
  NPC incidence rate will be compared between screening group and control group at 12-year follow-up.
Stage distribution at diagnosis for NPC patients by intervention group | December, 2019
  Stage distribution will be compared between screening group and control group at 12-year follow-up.
NPC overall survival by cases from the two intervention groups | December, 2019
  Survival rate will be compared between screening group and control group at 12-year follow-up.
Cost-effectiveness | December, 2019
  Cost-effectiveness of this screening program will be calculated at 12-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Minghuang Hong, M.D, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sihui Cancer Institute, Sihui, Guangdong
  - Cancer Research Institute of Zhongshan City, Zhongshan, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen WJ, Yu X, Lu YQ, Pfeiffer RM, Ling W, Xie SH, Wu ZC, Li XQ, Fan YY, Wu BH, Wei KR, Rao HL, Huang QH, Guo X, Sun Y, Ma J, Liu Q, Hildesheim A, Hong MH, Zeng YX, Ji MF, Liu Z, Cao SM. Impact of an Epstein-Barr Virus Serology-Based Screening Program on Nasopharyngeal Carcinoma Mortality: A Cluster-Randomized Controlled Trial. J Clin Oncol. 2025 Jan;43(1):22-31. doi: 10.1200/JCO.23.01296. Epub 2024 Oct 1. PMID 39353160
- [Derived] Ji MF, Sheng W, Cheng WM, Ng MH, Wu BH, Yu X, Wei KR, Li FG, Lian SF, Wang PP, Quan W, Deng L, Li XH, Liu XD, Xie YL, Huang SJ, Ge SX, Huang SL, Liang XJ, He SM, Huang HW, Xia SL, Ng PS, Chen HL, Xie SH, Liu Q, Hong MH, Ma J, Yuan Y, Xia NS, Zhang J, Cao SM. Incidence and mortality of nasopharyngeal carcinoma: interim analysis of a cluster randomized controlled screening trial (PRO-NPC-001) in southern China. Ann Oncol. 2019 Oct 1;30(10):1630-1637. doi: 10.1093/annonc/mdz231. PMID 31373615
- [Derived] Liu Z, Ji MF, Huang QH, Fang F, Liu Q, Jia WH, Guo X, Xie SH, Chen F, Liu Y, Mo HY, Liu WL, Yu YL, Cheng WM, Yang YY, Wu BH, Wei KR, Ling W, Lin X, Lin EH, Ye W, Hong MH, Zeng YX, Cao SM. Two Epstein-Barr virus-related serologic antibody tests in nasopharyngeal carcinoma screening: results from the initial phase of a cluster randomized controlled trial in Southern China. Am J Epidemiol. 2013 Feb 1;177(3):242-50. doi: 10.1093/aje/kws404. Epub 2012 Dec 19. PMID 23255783